CLINICAL TRIAL: NCT04954157
Title: Studies to Determine Whether Oxygen Sensing is Impaired in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-0898
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Hypoxia; SARS-CoV-2 Acute Respiratory Disease; Carotid Bodies
MeSH Terms: conditions — Hypoxia | interventions — Walk Test

STUDY DESIGN:
Intervention Model Description: Each group of subjects will be required to perform the same test, depending on what phase of the study they are recruited into. If the subject currently has been diagnosed with COVID-19 and fits all other criteria, they will be placed in the COVID-19 group. If the subject has not been diagnosed with COVID-19 and are considered healthy at that time, they will be placed on the healthy group.
Masking Description: There is no masking taking place in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Placebo Comparator): This arm will consist of health subjects, not infected with COVID-19
  Interventions: Diagnostic Test: Phase-1: Breath Holding Test; Diagnostic Test: Phase 2: 6-Minute Walk Test (6MWT)
- COVID 19 Subjects (Active Comparator): This arm will consist of subjects who are currently diagnosed with COVID-19 and fit all other criteria to be enrolled in this study.
  Interventions: Diagnostic Test: Phase-1: Breath Holding Test; Diagnostic Test: Phase 2: 6-Minute Walk Test (6MWT)

INTERVENTIONS:
Diagnostic Test: Phase-1: Breath Holding Test — In this phase of the study, each subject will be asked to hold their breath for up to 60 seconds or until they can longer hold it. While they are holding their breath, subjects will be hooked up to a monitor that will measure their Peripheral oxygen saturation (SpO2) respiratory rate (RR), and heart rate (HR).
Diagnostic Test: Phase 2: 6-Minute Walk Test (6MWT) — In this phase of the study, each subject will be asked to walk for 6 minutes in their hospital room or hallway. Their rate of perceived exertion will be measured while also hooked up to a monitor that will measure their Peripheral oxygen saturation (SpO2) respiratory rate (RR), and heart rate (HR).

SUMMARY:
The two-part phases will each have a unique patient population, The goal in this application is to see if that carotid bodies are "offline" is correct and to determine whether a cohort of SARS-Cov-2 patients can be identified who fit this profile and would be suitable for drug treatment.

The testing will require one group of subjects to hold their breaths for a short period while the investigators monitor vital signs and blood O2 levels. A second group of "healthier" COVID subjects will be asked perform a walk-test inside their rooms for six minutes while vital signs are monitored as well as blood O2 levels. If the subjects are in the healthy control group, they will perform the walk test in a designated hallway at the medical center also while there vitals are being monitored. The goal, using a mild stimulus, is to determine whether respiration increases if blood O2 saturation is decreased. If it does not, that would indicate a failure of the carotid body oxygen sensing system.

DETAILED DESCRIPTION:
Many patients infected with SARS-CoV-2 are hypoxic (O2 blood saturation below 92%). Many do not even realize they are hypoxic, since breathing can remain comfortable. In these patients, the normal physiologic responses to low oxygen, increased respiration, appears to be absent (Couzin-Frankel, 2020).

A wide variety of cell types within the body express the ACE2 receptor that is required by the virus to infect cells. This included the cells of the carotid body, which are the O2 sensors of the body. The investigators hypothesize that glomus cells of the carotid body are among the first cells infected due to their extremely high blood perfusion rates. After infection, they are "offline" and the body no longer recognizes that it is hypoxic. This can be extremely detrimental to patients that may require mechanical ventilation to re-establish normal blood O2 levels (>95% saturation). Death rates on patients using mechanical ventilators are very high and every effort should be made to keep patients off these machines.

Interestingly, hypoxia appears to be a common condition in SARS-CoV-2 infected people, with some showing serious respiratory conditions (acute respiratory distress syndrome - ARDS), but others not. The majority appear to die from a "cytokine storm", a massive reaction to the infection by the immune system (Xie et al., 2020). But many others are hypoxic and sick. Many medical centers are treating SARS-Cov-2 patients identically, placing them on mechanical respirators. Below is a short description from a German group from an editorial that was recently published (Gattinoni et al., 2020) suggesting that not all SARS-CoV-2 hypoxic patients are the same and so should not be treated identically.

It has been known for a long time that mechanical ventilation in ICU patients, not related to SARS-CoV-2, can be very hard on patients with death rates above 50% (Fialkow et al., 2014) and with very long recovery times (Griffiths & Jones, 1999). Patients admitted to ICUs who need mechanical ventilation are expected to have higher mortality rates compared with those who do not require respiratory support (Vincent et al., 2002) as a consequence of ventilator-induced lung injury (VILI). Intubated patients infected with SARS-CoV-2 also have very high death rates (Richardson et al., 2020). Undoubtedly, they are the sickest of the sick. Nonetheless, everything possible should be done to prevent intubation a policy consistent with University of Chicago usage of high flow nasal cannulation. The investigators goal with this IRB submission is to identify a cohort of SARS-CoV-2 patients that are hypoxic but their breathing is not responding correctly to the hypoxia ("silent hypoxia"). It is possible that these patients can be treated with drugs, in order to keep them from intubation for as long as possible.

Phase I - Study of silent hypoxia in SARS-CoV-2 infected patients. Phase 1 will recruit 40 subjects with documented SARS-CoV-2 infection and another 40 healthy subjects as the control group. Totaling 80 subjects in the first phase. This large a group is not required to determine if "silent hypoxia" exists, rather to determine the percentage of patients exhibiting altered oxygen sensing, among this patient population.

This Phase will include observation and collection of clinical data that is routinely captured in hospitalized COVID patients. All COVID-19 patients at the University of Chicago Medical Center (UCMC) are connected to telemetry monitors that measure vital signs. Peripheral oxygen saturation (SpO2), respiratory rate (RR), and heart rate (HR) are continuously measured by the telemetry monitors. Blood pressure is intermittently checked and measured by the telemetry monitor at an interval determined by physician orders at admission.

Prior to the subject's performing the test, they will have the option of watching a brief instructional video, created by the PI, on how to correctly perform the phase one test. Both the COVID and healthy subjects will have this option, if they feel they need further instruction other than what the clinician administering the test has already provided. Once the subject feels ready, will then be asked to hold their breaths up to 60 seconds or until they can no longer hold their breath. Every patient will be asked to hold their breath 3 times with 5 minutes of rest between trials. Subjects will be instructed to hold their breath and their vital signs will be recorded before, during, and after breath holding by the patient's attending physician in the COVID unit. The goal is to see whether breath holding makes the subject uncomfortable, as it would do in a normal subject. If their O2 sensing is impaired the drive to breath may be absent or diminished. After the breath holding stops, it is expected that the patient may start to gasp and breathe more rapidly, to make up for the oxygen deficit. Will all subjects respond to hypoxia correctly? Or will some subjects ignore the hypoxia, because they do not know they need to stop? In that case, a member of the study team will stop them.

To ensure patient safety the attending physicians will instruct and monitor subjects while they are participating in this study. Changes in O2 saturation below 85% or an absolute drop of more than 8% will trigger the physician to instruct the patient to start breathing. Table 1, below, will guide breath-holding criteria.

Phase II - Studies of silent hypoxia in SARS-CoV-2 infected patients. Phase 2 will recruit 10 subjects and ask them ambulate for six minutes in their hospital room. This length of time is adapted from the six minute walk test (6MWT), which is a well validated measure of both aerobic and functional capacity (Troosters et al., 2002; Enright, 2003). The purpose of the experiment is to test whether simple physical exertion in ambulatory COVID patients is associated with reductions in SpO2 and/or physiologic changes in vital signs. The 6MWT will be adapted and ask subjects to ambulate back and forth in their room (rather than along a 100m corridor), since this study is primarily interested in the physiologic responses to exertion (rather than total distance walked). The study team will also measure at baseline and after completion of walking a set of vital signs as well as ask subjects about their perceived exertion using the Borg Rating of Perceived exertion instrument. In this phase, patients will be instructed and continuously monitored by attending physicians working in the COVID unit. The attending physicians will monitor these patients by standing outside of the patient's room but in full view of the patient through the window and/or doorway in the COVID unit.

For this phase, patients will be recruited with a documented AM-PAC score ≥19. The AM-PAC score is documented daily by UCMC nurses in the nursing and therapy flow sheets within EPIC. The score of ≥19 is used by both UCMC nurses and physical therapists to indicate patients' functional independence. The daily AM-PAC scoring of patients by nurses at UCMC is required and based on an adapted version of the Activity Measure for Post-Acute Care (AM-PAC) instrument (Haley et al., 2004). This nursing requirement and the adapted AM-PAC scoring was a joint UCMC nursing and physical therapy initiative, Project Walk, to better target patients who may or may not need PT during their admission based on their functional mobility.

To ensure patient safety the attending physicians will instruct and monitor patients while they are participating in this study. Changes in O2 saturation below 85% or an absolute drop of more than 5% will trigger the physician to instruct the patient to start breathing.

What if all SARS-CoV-2 patients have impaired O2 sensing? This may not be out of the question, since it appears that loss of smell and taste are reliable indicators of infection (Menni et al.). In that case, the investigators population studies will indicate that everyone is hypoxic when stressed.

Subject Identification, Recruitment & Payment All COVID subjects will be recruited and enrolled from the COVID unit at the University of Chicago Medical Center (UCMC). The healthy subjects will come from the faculty and staff from UCMC. To avoid any possible bias, healthy volunteers will not have any relationship to this study prior or be under the supervision of the investigators at the time they participate in this study. The healthy subjects will not be hospitalized at the time they are recruited for this study. Subjects will not be compensated for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* We intend to include patients who meet the following criteria in the study.

  * Anyone with COVID 19 positive
  * Willing to give consent for the study.
  * 18 years of age and up
  * A documented AM-PAC score>19 (Phase II Only)

Exclusion Criteria:

* We plan to exclude patients who meet any of the following criteria:

  * Patients that cannot walk safely
  * Non-English Speakers
  * Covid 19 patients who requires intubation or HFNC (high flow nasal cannula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Determine whether COVID 19 impairs the function of oxygen sensors in carotid bodies by utilizing the breath hold test. | 1 Day
  This will determined by asking subjects to take a regular breath, and exhale, hold it until you have to take another breath or until 1) you cannot hold it anymore; 2) up to 60 sec; 3) your O2 saturation falls to 85% or lower, 4) you feel dizzy, or 5) heart rate change > 30 % of the baseline (pre breath holding heart rate.
Determine whether COVID 19 impairs the function of oxygen sensors in carotid bodies by utilizing the 6-Minute Walk Test | 1 Day
  To determine and report six-minute walk test performance, assessing the rate of exertion for each subject by using the Borg Rating of Perceived exertion instrument. This scale is from 6 to 20, where 6 means "No exertion at all" and 20 means "Maximal exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng (Jimmy) Xie, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No